CLINICAL TRIAL: NCT02393027
Title: Quantification of Dopamine Active Transporter (DAT) in Humans: Validation of a New Radiophamaceutical, the [18F] LBT-999
Acronym: LBT 999
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enough inclusions for interpretation
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO14-MJR / LBT-999
Record Dates: First submitted 2015-03-06; First posted 2015-03-19 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients (Experimental): 10 idopathic parkinson disease
  Interventions: Drug: [18F] LBT-999 PET
- controls subjects (Active Comparator): 10 healthy controls (no parkinson disease)
  Interventions: Drug: [18F] LBT-999 PET

INTERVENTIONS:
Drug: [18F] LBT-999 PET

SUMMARY:
Idiopathic Parkinson's disease (IPD) is a degenerative disease affecting the dopaminergic system. Clinical symptoms of IPD commonly begin after the loss of at least 40 to 50% of striatal dopaminergic terminals (specially putaminal terminals).

The Dopamine neuronal transporter (DAT) is a highly expressed protein in the membrane of presynaptic nigrostriatal dopaminergic terminals. The use of a DAT's radioligand in the initial stages of the disease would lead to an early detection of nigral cell loss.

Currently, only one DAT's radioligand has obtained marketing authorization in France, the 123I-FPCIT, for use in Single Photon Emission Computed Tomography (SPECT).

Otherwise, the Positron Emission Tomography (PET), a more sensitive technology than SPECT with higher resolution has become for a few years the new gold standard for visual analysis and quantification of neurotransmission systems (including the dopaminergic system).

A DAT tracer labelled with Carbon 11 ([11C] PE2l) have been developed and is currently used as a reference in various research centers.

However, in order to enable a clinical use of this tracer (which currently can't be because of the too short period of Carbon 11), the unit INSERM U930 "Imaging and Brain" in collaboration with the CERRP (Center for Studies and Research on Radiopharmaceuticals) developed a new version of this tracer, labelled with 18-fluor: the [18F] LBT-999.

The main goal of this study is to compare the [18F] LBT-999 uptake between a group of patients suffering from a Parkinsonien syndrome to a group healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Criteria common to all participants:

* Age between 45 and 75 years old
* Signed informed consent
* Affiliated to a social security system

Criteria for patients:

* idiopathic Parkinson's disease according to the UKPDSBB criteria
* stage 1-3 Hoen and Yahr (unilateral disease to moderate or mild bilateral disease in a self patient )

Criteria for healthy volunteers:

* matching according to age (± 5 years)

Exclusion Criteria:

Criteria common to all participants:

* history of taking an antipsychotic or any other drug with a dopaminergic effect in the previous 6 months
* contraindications to MRI
* person with severe claustrophobia
* patient with a legal protection measure
* alcohol or drug abuse history (in the past 10 years)
* history of progressive disease that can affect the central nervous system (blood pressure greater than or equal to 180/100 mmHg, chronic lung disease with hypoxia, heart failure stage 4)
* all medical and surgical affection older than 3 months
* history of stroke
* history of head trauma (coma> 24h)
* MMS<24
* pregnancy or lactating woman without reliable contraception

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Binding potential of [18F] LBT-999 | one year

SECONDARY OUTCOMES:
DAT striatal density by estimating the LBT-999 distribution volume | one year
presence of lipophilic metabolites | one year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Tours, France

REFERENCES:
- [Background] Agid Y. Parkinson's disease: pathophysiology. Lancet. 1991 Jun 1;337(8753):1321-4. doi: 10.1016/0140-6736(91)92989-f. No abstract available. PMID 1674304
- [Background] Brooks DJ, Pavese N. Imaging biomarkers in Parkinson's disease. Prog Neurobiol. 2011 Dec;95(4):614-28. doi: 10.1016/j.pneurobio.2011.08.009. Epub 2011 Aug 30. PMID 21896306
- [Background] Brooks DJ. Imaging dopamine transporters in Parkinson's disease. Biomark Med. 2010 Oct;4(5):651-60. doi: 10.2217/bmm.10.86. PMID 20945978
- [Background] Chalon S, Hall H, Saba W, Garreau L, Dolle F, Halldin C, Emond P, Bottlaender M, Deloye JB, Helfenbein J, Madelmont JC, Bodard S, Mincheva Z, Besnard JC, Guilloteau D. Pharmacological characterization of (E)-N-(4-fluorobut-2-enyl)-2beta-carbomethoxy-3beta-(4'-tolyl)nortropane (LBT-999) as a highly promising fluorinated ligand for the dopamine transporter. J Pharmacol Exp Ther. 2006 Apr;317(1):147-52. doi: 10.1124/jpet.105.096792. Epub 2005 Dec 9. PMID 16339913
- [Background] de Rijk MC, Tzourio C, Breteler MM, Dartigues JF, Amaducci L, Lopez-Pousa S, Manubens-Bertran JM, Alperovitch A, Rocca WA. Prevalence of parkinsonism and Parkinson's disease in Europe: the EUROPARKINSON Collaborative Study. European Community Concerted Action on the Epidemiology of Parkinson's disease. J Neurol Neurosurg Psychiatry. 1997 Jan;62(1):10-5. doi: 10.1136/jnnp.62.1.10. PMID 9010393
- [Background] Fernagut PO, Li Q, Dovero S, Chan P, Wu T, Ravenscroft P, Hill M, Chen Z, Bezard E. Dopamine transporter binding is unaffected by L-DOPA administration in normal and MPTP-treated monkeys. PLoS One. 2010 Nov 22;5(11):e14053. doi: 10.1371/journal.pone.0014053. PMID 21124922
- [Background] Hsiao IT, Weng YH, Lin WY, Hsieh CJ, Wey SP, Yen TC, Kung MP, Lu CS, Lin KJ. Comparison of 99mTc-TRODAT-1 SPECT and 18 F-AV-133 PET imaging in healthy controls and Parkinson's disease patients. Nucl Med Biol. 2014 Apr;41(4):322-9. doi: 10.1016/j.nucmedbio.2013.12.017. Epub 2014 Jan 10. PMID 24503330
- [Background] Serriere S, Tauber C, Vercouillie J, Guilloteau D, Deloye JB, Garreau L, Galineau L, Chalon S. In vivo PET quantification of the dopamine transporter in rat brain with [(1)(8)F]LBT-999. Nucl Med Biol. 2014 Jan;41(1):106-13. doi: 10.1016/j.nucmedbio.2013.09.007. Epub 2013 Oct 8. PMID 24210285
- [Background] Schillaci O, Pierantozzi M, Filippi L, Manni C, Brusa L, Danieli R, Bernardi G, Simonetti G, Stanzione P. The effect of levodopa therapy on dopamine transporter SPECT imaging with( 123)I-FP-CIT in patients with Parkinson's disease. Eur J Nucl Med Mol Imaging. 2005 Dec;32(12):1452-6. doi: 10.1007/s00259-005-1922-9. Epub 2005 Sep 8. PMID 16151764
- [Background] Sharma S, Moon CS, Khogali A, Haidous A, Chabenne A, Ojo C, Jelebinkov M, Kurdi Y, Ebadi M. Biomarkers in Parkinson's disease (recent update). Neurochem Int. 2013 Sep;63(3):201-29. doi: 10.1016/j.neuint.2013.06.005. Epub 2013 Jun 19. PMID 23791710
- [Background] Snow BJ, Tooyama I, McGeer EG, Yamada T, Calne DB, Takahashi H, Kimura H. Human positron emission tomographic [18F]fluorodopa studies correlate with dopamine cell counts and levels. Ann Neurol. 1993 Sep;34(3):324-30. doi: 10.1002/ana.410340304. PMID 8363349
- [Background] Varrone A, Stepanov V, Nakao R, Toth M, Gulyas B, Emond P, Deloye JB, Vercouillie J, Stabin MG, Jonsson C, Guilloteau D, Halldin C. Imaging of the striatal and extrastriatal dopamine transporter with (18)F-LBT-999: quantification, biodistribution, and radiation dosimetry in nonhuman primates. J Nucl Med. 2011 Aug;52(8):1313-21. doi: 10.2967/jnumed.111.089953. Epub 2011 Jul 15. PMID 21764797